CLINICAL TRIAL: NCT07083700
Title: The Impact of the Frame™ Platform on Infertility Patient Retention and Emotional Health: A Randomized Controlled Pilot Study
Brief Title: Frame Support Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inception Fertility Research Institute, LLC (Industry)
Collaborators: Reframe Health, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRI-RH-2025-001
Record Dates: First submitted 2025-06-24; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Fertility Issues; Emotional Stress
MeSH Terms: conditions — Infertility; Stress, Psychological

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention)
- Frame Access (Experimental)
  Interventions: Behavioral: Frame Access

INTERVENTIONS:
Behavioral: Frame Access — FRAME™ provides a collaborative care platform that connects patients with evidence-based resources, education and support from a dedicated care team throughout their reproductive health care journey. More specifically, for patients exploring fertility treatment. Frame supplements the patient experience by providing patients with direct contact to board-certified fertility coaches and resources that can be accessed between appointments in a web-based application. Regular use of Frame's platform may help patients make lifestyle changes that can improve their fertility outcomes as well as boost their emotional health throughout the treatment process and reduce feelings of overwhelm and loneliness which can lead to patients dropping out of care.
  Arms: Frame Access

SUMMARY:
This is a randomized, controlled pilot study evaluating an intervention of non-significant risk. Potential subjects will be women who have completed an initial new patient consultation at one of the participating fertility clinics. Approximately 400 subjects will be enrolled from multiple fertility clinics.

DETAILED DESCRIPTION:
All participants will complete a psychological questionnaire at enrollment. The questionnaire will include the Perceived Stress Scale (PSS), the Personal Health Questionnaire Depression Scale (PHQ-8), and the Copenhagen Multi-Centre Psychosocial Infertility- Fertility Problem Stress Scale (COMPI-FPSS). Participants will then be randomized 1:1 to the control group or intervention group. Participants in the control group will not be asked to take any additional action for six months. Participants in the intervention group will be given access to FRAME which will provide them with resources and an external care team to utilize during their fertility care. The intervention group is encouraged to use FRAME and its resources for six months. After six months, participants in both groups will complete a post-study psychological questionnaire. Data will be collected from medical records of all participants for up to nine months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Participants have completed a new patient consult at one of the participating fertility clinics
* Participants must be able to read, write and speak English
* Participants must have access to a smart phone and internet connection

Exclusion Criteria:

* Patients who are currently using a fertility coach (in-person, remote, or online)
* Patients planning egg freezing only
* Patients who have received treatment at another fertility center
* Patients planning egg donation
* Patients currently participating in another clinical trial or study involving an intervention.

Ages: 22 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This research is targeting patients who are the primary recipient of fertility treatment.
Enrollment: 400 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Fertility treatment initiation | This will be evaluated at the end of patient's study participation, approximately 6 months post enrollment.
  To observe whether the patient started fertility treatment.

SECONDARY OUTCOMES:
Time to fertility treatment initiation | This will be evaluated at the end of patient's study participation, approximately 6 months post enrollment.
  To observe the interval between study enrollment and start fertility treatment, if any.

OTHER OUTCOMES:
Patient Health Questionnaire (PHQ-8) | From enrollment to six months after enrollment
  Patients will complete the Patient Health Questionnaire (PHQ-8) for depression screening at baseline and end of study. Scores of 10 and above suggest the presence of Major Depressive Disorder with higher scores being more severe.
Copenhagen Multi-Centre Psychosocial Infertility- Fertility Problem Stress Scale (COMPI-FPSS) | From enrollment to 6 months after enrollment.
  Patients will complete the Copenhagen Multi-Centre Psychosocial Infertility- Fertility Problem Stress Scale (COMPI-FPSS) at baseline and end of study. Lower scores indicate lower stress.
Perceived Stress Scale (PSS-10) | From enrollment to 6 months after enrollment.
  Patients will complete the Perceived Stress Scale (PSS-10) at baseline and end of study. Scores will be interpreted as 0-13: Low stress; 14-26: Moderate stress; 27-40: High perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Inception Fertility Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No